CLINICAL TRIAL: NCT06945718
Title: Prospective Trials on Clinical Outcomes of Indocyanine Green Tracer Using in Laparoscopic Gastrectomy With D2 Extra-regional Lymph Node Dissection for Locally Advanced Gastric Cancer (FUGES-30)
Brief Title: Clinical Outcomes of Indocyanine Green Tracer Using in Laparoscopic Gastrectomy With Extended Lymphadenectomy Beyond D2 for Locally Advanced Gastric Cancer (FUGES-30)
Status: Recruiting | Type: Observational
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Chief doctor, phD, FACS, Fujian Medical University
Other Study IDs: FUGES-30
Record Dates: First submitted 2025-03-21; First posted 2025-04-25 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Gastric Cancer; Surgery
Keywords: Gastric Cancer; Laparoscopic Gastrectomy; Indocyanine Green Tracer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- laparoscopic gastrectomy with beyond D2 regional fluorescent lymph node dissection with ICG group: ICG with D2+ group
  Interventions: Procedure: beyond D2 regional lymph node dissection
- laparoscopic gastrectomy with D2 regional lymph node dissection with ICG group: ICG with D2 group
  Interventions: Procedure: beyond D2 regional lymph node dissection

INTERVENTIONS:
Procedure: beyond D2 regional lymph node dissection — dissect the lymph nodes outside the extent of D2 LN region.

SUMMARY:
Taking patients with locally advanced gastric adenocarcinoma (cT2-4a, N-/+, M0) as the research subjects, to evaluate whether the clinical efficacy of laparoscopic beyond D2 regional lymph node dissection for gastric cancer with indocyanine green tracer is better or not.

ELIGIBILITY:
Inclusion Criteria:

Age from 18 to 75 years Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy cT2-4a, N-/+, M0 at preoperative evaluation according to the AJCC Cancer Staging Manual, 8th Edition No distant metastasis, no direct invasion of pancreas, spleen or other adjacent organs in the preoperative examinations Performance status of 0 or 1 on the ECOG (Eastern Cooperative Oncology Group) scale ASA (American Society of Anesthesiology) class I to III Written informed consent

Exclusion Criteria:

Women during pregnancy or breast-feeding Severe mental disorder History of previous upper abdominal surgery (except for laparoscopic cholecystectomy) History of previous gastric surgery (including ESD/EMR for gastric cancer) Enlarged or bulky regional lymph node (diameter over 3cm) supported by preoperative imaging including enlarged or bulky lymph nodes in D3 region.

Other malignant disease within the past 5 years History of unstable angina or myocardial infarction within past six months History of cerebrovascular accident within past six months History of continuous systematic administration of corticosteroids within one month Requirement for simultaneous surgery for other disease Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer FEV1 (forced expiratory volume in one second)<50% of predicted values Diffuse invasive gastric cancer Tumors preoperatively confirmed to involve the squamocolumnar junction or duodenum History of an iodine allergy Patients who declined laparoscopic surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age from 18 to 75 years Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy cT2-4a, N-/+, M0 at preoperative evaluation according to the AJCC Cancer Staging Manual, 8th Edition
Sampling Method: Non-Probability Sample
Enrollment: 760 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival rate | 3 years
  Disease-free survival is calculated from the day of surgery to the day of recurrence or death

SECONDARY OUTCOMES:
Total number of retrieved lymph nodes | 30 days
  Total number of retrieved lymph nodes
Noncompliance rate of lymph node dissection | 30 days
  The LN dissection rate was determined by the number of patients in whom a LN station was harvested divided by the total number of patients who required retrieval at the corresponding LN station. Within the scope of D2 dissection, LN noncompliance was defined as the absence of LNs that should have been resected from > 1 LN station.
Relationship between fluorescent lymph nodes in group A and total number of lymph nodes in group A | 30 days
  Relationship between the number of fluorescent lymph nodes in group A and total number of lymph nodes in group A
Relationship between fluorescent lymph nodes in Group A and positive lymph nodes in Group A (positive rate) | 30 days
  The number of positive lymph nodes in fluorescent lymph nodes is divided by the number of total fluorescent lymph nodes in Group A (True positive rate).
Relationship between fluorescent lymph nodes in Group A and negative lymph nodes in Group A (false positive rate) | 30 days
  The number of negative lymph nodes in fluorescent lymph nodes is divided by the number of total fluorescent lymph nodes in Group A (false positive rate).
Relationship between non-fluorescent lymph nodes in Group A and negative lymph nodes in group A (negative rate) | 30 days
  The number of negative lymph nodes in not fluorescent lymph nodes is divided by the number of total not fluorescent lymph nodes in group A (True negative rate).
Relationship between nonfluorescent lymph nodes in Group A and positive lymph nodes in Group A (false negative rate) | 30 days
  The number of positive lymph nodes in not fluorescent lymph nodes is divided by the number of total not fluorescent lymph nodes in Group A (false negative rate).
Relationship between fluorescent lymph nodes in group B and total number of lymph nodes in group B | 30 days
  Relationship between the number of fluorescent lymph nodes in group B and total number of lymph nodes in group B
Relationship between fluorescent lymph nodes in Group B and positive lymph nodes in Group B (positive rate) | 30 days
  The number of positive lymph nodes in fluorescent lymph nodes is divided by the number of total fluorescent lymph nodes in Group B (True positive rate).
Relationship between fluorescent lymph nodes in Group B and negative lymph nodes in Group B (false positive rate) | 30 days
  The number of negative lymph nodes in fluorescent lymph nodes is divided by the number of total fluorescent lymph nodes in Group A (false positive rate).
Relationship between non-fluorescent lymph nodes in Group B and negative lymph nodes in group B (negative rate) | 30 days
  The number of negative lymph nodes in not fluorescent lymph nodes is divided by the number of total not fluorescent lymph nodes in group B (True negative rate).
Relationship between nonfluorescent lymph nodes in Group B and positive lymph nodes in Group B (false negative rate) | 30 days
  The number of positive lymph nodes in not fluorescent lymph nodes is divided by the number of total not fluorescent lymph nodes in Group B (false negative rate).
Number of metastatic lymph nodes | 30 days
  Number of metastatic lymph nodes
Metastasis rate of lymph nodes | 30 days
  Metastasis rate of lymph nodes
Postoperative complications | 30 days
  Postoperative complications were evaluated within 30 days following surgery. These postoperative complications include gastrointestinal-related complications, incision-related complications, respiratory complications, cardiovascular and cerebrovascular complications, urinary system complications, infection complications, embolism complications, and other complications. The grading of postoperative complications adopts the Clavien-Dindo classification.
Mortality rates | 30 days
  Patient died during hospitalization.
3-year overall survival rate | 3 years
  3-year overall survival rate
3-year recurrence pattern | 3 years
  3-year recurrence pattern
Postoperative recovery course | 30 days
  Time to first flatus after surgery, time to first ambulation after surgery, time to first liquid diet after surgery, time to first semi-liquid diet after surgery, length of hospital stay after surgery.
The incidence of intraoperative complications | 30 days
  Intraoperative complications were defined as bleeding due to named vessel injury, injury to visceral organs, mechanical factor-related problems, cardiopulmonary dysfunction due to hypercapnia, and other complications
Inflammatory and immune response | 7 days
  the values of hemoglobin, prealbumin, albumin, C-reactive protein, and white blood cell count from peripheral blood before the operation and on postoperative day 1, 3, 5 are recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Ming Huang, Prof., Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No